CLINICAL TRIAL: NCT06134596
Title: Correlation of Clitoral Hood and Labia Minora Measurements and Female Genital Self Image Scale (FGSIS) Scores in Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Evrim Ebru Kovalak, Medical doctor, Bagcilar Training and Research Hospital
Other Study IDs: 2023-06-06
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Genital Diseases, Female; Vulva
Keywords: Genital diseases, vulva
MeSH Terms: conditions — Genital Diseases, Female; Genital Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the relationship between women's labium minora and clitoral hood measurements and Female Genital Self Image Scale (FGSIS) scores.

DETAILED DESCRIPTION:
The main purpose of our study is to measure the labium minora and clitoral hood in women who apply to our clinic with gynecological disorders, evaluate them with FGSIS (Female Genital Self Image Scale) scores, and look at the relationship between genital area perception and labium minora and clitoral hood dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Women who apply for outpatient gynecological control, are between the ages of 18-45, are sexually active, do not have additional endocrinological or malignant diseases, and are not pregnant or in menopause.

Exclusion Criteria:

* Those who are not sexually active, have varying degrees of pelvic organ prolapse or urinary incontinence, have a malignancy, or have an endocrinological disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women who apply for outpatient gynecological control, are between the ages of 18-45, are sexually active, do not have additional endocrinological or malignant diseases, and are not pregnant or in menopause.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of genital measurement with genital perception | 2 months
  Since the genital aesthetic trend is very popular today, it is important to understand the importance of labia minora and clitoral hood measurements in female genital perception.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Ebru Kovalak, MD, Principal Investigator — Bagcilar Training and Research Hospital
Locations (1):
- Bagcilar Teaching and Research Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Widschwendter A, Riedl D, Freidhager K, Abdel Azim S, Jerabek-Klestil S, D'Costa E, Fessler S, Ciresa-Konig A, Marth C, Bottcher B. Perception of Labial Size and Objective Measurements-Is There a Correlation? A Cross-Sectional Study in a Cohort Not Seeking Labiaplasty. J Sex Med. 2020 Mar;17(3):461-469. doi: 10.1016/j.jsxm.2019.11.272. Epub 2020 Jan 7. PMID 31918983